CLINICAL TRIAL: NCT05576857
Title: The Effects of Neck Hyperextension on Neck Blood Flow, Cerebral Oximetry and Cognitive Functions in Adult Healthy Volunteers
Brief Title: Effects of Cervical Hyperextension on Cervical Blood Flow, Cerebral Oximetry and Cognitive Functions.
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Other Study IDs: drozlemersoy2
Record Dates: First submitted 2022-10-07; First posted 2022-10-13 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Hyperextension Injury of Neck
Keywords: hyperextension of neck; cervical blood flow; cerebral oxygen saturation; optic nerve sheath
MeSH Terms: interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Doppler ultrasonography — All volunteers will be monitored with cerebral oximeter, asked to answer the Montreal cognitive assessment test and cervical blood flow values and optic nerve sheath diameter will be determined with Doppler ultrasonography.
  Other Names: Montreal cognitive assessment test; cerebral oximeter

SUMMARY:
The goal of this observational study is to determine the effects of cervical hyperextension on cerebral oximetry and cognitive functions in healthy individuals without other additional factors such as anesthesia and surgical stress. The main questions it aims to answer are:

* Can cervical hyperextension cause changes in cerebral oxygenation in non-anesthetized healthy individuals?
* Can cervical hyperextension cause changes in cervical and cerebral blood flow in non-anesthetized healthy individuals?
* Can cervical hyperextension cause changes in cognitive functions in non-anesthetized healthy individuals?
* Can cervical hyperextension cause changes in optic nerve sheath diameter in non-anesthetized healthy individuals? Participants will be monitored with cerebral oximeter device and asked to answer Montreal cognitive function test before and during cervical hyperextension position. The researchers will evaluate the changes in cervical and cerebral blood flow ultrasonographically before and during cervical hyperextension position.

DETAILED DESCRIPTION:
Some operations are performed in the cervical hyperextension position. During the cervical hyperextension position, changes in neck blood flow as a result of stretching of neck vessels can occur. These changes can be observed as an increase or decrease in cerebral blood flow. Changes in cerebral blood flow can lead to changes in brain oxygenation and affect cognitive functions.

Aim: This study aims to show the effects of cervical hyperextension on cerebral oximetry and cognitive functions in healthy individuals without other additional factors such as anesthesia and surgical stress.

Method: Healthy volunteers who meet the specified criteria and sign informed consent will be included in the study. All volunteers will be asked to answer validated Montreal cognitive assessment test in Turkish. Cerebral oximetry will be monitored by 2 probes placed on the frontal bone while all volunteers are lying in a supine position with the neck in a neutral position. Basal cerebral oximetry values will be recorded. In the same position cervical blood flow values and optic nerve sheath diameter will be measured by the same and experienced researcher non-invasively with a Doppler ultrasonography device and recorded. Optimum cervical hyperextension position will be obtained by placing the standard pad under the neck of the volunteers. In the meantime cerebral oximetry values will be recorded. Cervical blood flow will be re-measured in this position non-invasively with a Doppler ultrasonography device and recorded. Cerebral oximeter values will be recorded every 5 minutes for 30 minutes. In the end of 30 minutes period of hyperextension position the cervical blood flow and optic nerve sheath diameter will be measured again non-invasively with a Doppler ultrasonography device and recorded. Immediately afterwards, the Montreal cognitive assessment test will be repeated without changing the position. After all measurements are completed, the procedure will be terminated by resting the volunteer in neutral position for 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years, healthy volunteers

Exclusion Criteria:

* diabetes mellitus,
* chronic obstructive pulmonary disease,
* Liver failure,
* Kidney failure,
* Past coronary arteria by-pass graft history,
* Hemoglobinopathies,
* Anemia,
* hypertensive patients,
* Alzheimer's disease,
* neurodegenerative diseases,
* mental retardation,
* Vertebrobasilar system anomalies detected in magnetic resonance-angiography

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 55 healthy volunteers between age of 18-65 years who meet the specified criteria, agreed to participate and signed informed consent will be included in the study.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the cervical blood flow rates | Cervical blood flow measurement will be performed 3 times in 30 minute period.
  Cervical blood flow measurement will be performed 3 times by the same and experienced researcher with the same Doppler ultrasonography device; before cervical hyperextension in neutral position, in the first 5 minutes of cervical hyperextension, in the end of 30 minutes period of cervical hyperextension position.
Change from baseline in the optic nerve sheath diameter | Optic nerve sheath diameter measurement will be performed 3 times in 30 minute period.
  Optic nerve sheath diameter measurement will be performed 2 times by the same and experienced researcher with the same Doppler ultrasonography device:
  before cervical hyperextension in neutral position, in the end of 30 minutes period of cervical hyperextension position.
Change from baseline in the cerebral oximeter values | Cerebral oxygenisation values will be measured continuously before and during the cervical hyperextension position and recorded in every 5 minutes in 30 minute period.
  Cerebral oxygenisation values will be measured continuously before and during the cervical hyperextension position with a transcutaneous near infrared spectroscope device (NIRS) via two transcutaneous probes placed on the frontal bone non-invasively and recorded.
Change from baseline in the Montreal cognitive assessment test | Montreal cognitive assessment test will be performed 2 times in 30 minute period.
  All volunteers will be asked to answer the Montreal cognitive assessment test 2 times by the same researcher; before cervical hyperextension in neutral position, in the end of 30 minutes period of cervical hyperextension position.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ersoy Karka, Principal Investigator — Düzce University Faculty of Medicine
Locations (1):
- Duzce University Faculty of Medicine, Düzce, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided